CLINICAL TRIAL: NCT03036384
Title: Estimation of the ED95 of Intrathecal Hyperbaric Prilocaine 2% With Sufentanyl for Scheduled Cesarean Delivery : a Dose-finding Study Bases on the Continual Reassessment Method (CRM)
Brief Title: Estimation of the ED95 of Intrathecal Hyperbaric Prilocaine 2% With Sufentanyl for Scheduled Cesarean Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NB076201627436
Record Dates: First submitted 2017-01-12; First posted 2017-01-30 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Pregnant Women
Keywords: scheduled cesarean delivery; spinal anesthesia; local anesthesia
MeSH Terms: interventions — Sufentanil; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 : HB prilocaine 2%, 45mg (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2%; Drug: Sufentanil; Drug: Morphine
- Cohort 2 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 3 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 4 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 5 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 6 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 7 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 8 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 9 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine
- Cohort 10 : HB prilocaine 2%, (30-55mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2%, associated with sufentanyl, will be administrated at the dose initial of 45 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). Possible dose levels are 30, 35, 40, 45, 50, 55mg.
  Interventions: Drug: HB Prilocaine 2% (varying dose); Drug: Sufentanil; Drug: Morphine

INTERVENTIONS:
Drug: HB Prilocaine 2% (varying dose) — Varying dose of hyperbaric (HB) prilocaine 2% according to sensitive response of previous subjects. The dose of hyperbaric prilocaine 2% will be administrated intrathecally with 100µg of morphine and 2.5µg of sufentanyl
  Other Names: Tachipri
  Arms: Cohort 10 : HB prilocaine 2%, (30-55mg); Cohort 2 : HB prilocaine 2%, (30-55mg); Cohort 3 : HB prilocaine 2%, (30-55mg); Cohort 4 : HB prilocaine 2%, (30-55mg); Cohort 5 : HB prilocaine 2%, (30-55mg); Cohort 6 : HB prilocaine 2%, (30-55mg); Cohort 7 : HB prilocaine 2%, (30-55mg); Cohort 8 : HB prilocaine 2%, (30-55mg); Cohort 9 : HB prilocaine 2%, (30-55mg)
Drug: HB Prilocaine 2% — The dose of 45mg of hyperbaric (HB) prilocaine 2% will be administrated intrathecally with 100µg of morphine and 2.5µg of sufentanyl
  Other Names: Tachipri
  Arms: Cohort 1 : HB prilocaine 2%, 45mg
Drug: Sufentanil — 2.5µg sufentanyl
Drug: Morphine — 100 µg Morphine

SUMMARY:
Hyperbaric bupivacaine 0.5% associated with opioids is the local anesthetic the most commonly used for spinal injection in cesarean section. Nevertheless, its use often results in a long duration of motor nerve block and a haemodynamical instability. Recently developped, the Prilocaine, with its new 2% hyperbaric formulation, seems to offer a good alternative for hyperbaric bupivicaine. A first study has determined the ED95 of hyperbaric prilocaine 2% for intrathecal anesthesia in scheduled cesarean delivery. As opioid adjuvants potentiate the effect of the local anesthetics while decreasing their dose-related side effects, the aim of this study is to determine the ED95 of hyperbaric prilocaine 2% with sufentanyl for scheduled cesarean delivery under spinal anesthesia,by using the Continual Reassessment Method (CRM)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) < III
* Age 18-40 year
* Body Weight <100 kg
* Height between 155 and 175 cm
* Gestational age>37 SA
* Elective cesarean delivery
* Singleton pregnancy
* Non complicated pregnancy
* Signed informed consent obtained prior to any study specific assessments and procedures

Exclusion Criteria:

* Twin pregnancy
* History of 2 cesarean section or more
* Diabetes and gestational diabetes
* Placenta praevia
* Congenital foetal abnormality
* Patient in labour
* Membrane rupture
* Known allergy to local anaesthetics
* Disagreement of the patient
* Pregnancy-induced hypertension
* Pre eclampsia and eclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Philippe Goffard, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- University Hospital Saint-Pierre, Université Libre de Bruxelles (ULB), Brussels Capital Region, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Background] Gupta PK, Chevret S, Zohar S, Hopkins PM. What is the ED95 of prilocaine for femoral nerve block using ultrasound? Br J Anaesth. 2013 May;110(5):831-6. doi: 10.1093/bja/aes503. Epub 2013 Feb 7. PMID 23393153
- [Derived] Goffard P, Vercruysse Y, Leloup R, Fils JF, Chevret S, Kapessidou Y. Determination of the ED95 of intrathecal hyperbaric prilocaine with sufentanil for scheduled cesarean delivery: a dose-finding study based on the continual reassessment method. BMC Anesthesiol. 2020 Nov 26;20(1):293. doi: 10.1186/s12871-020-01199-0. PMID 33243149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at CHU Saint-Pierre.
Pre-assignment Details: Possible doses of HB prilocaine range from 30 to 55mg, but actual administrated doses will be defined by CRM
Groups:
- Cohort 1: 45mg HB prilocaine initial dose; 4 patients
- Cohort 2; Cohort 3: 40mg HB prilocaine following CRM results; 4 patients
- Cohort 4: 35mg HB prilocaine following CRM results; 4 patients
- Cohort 5: 50mg HB prilocaine following CRM results, 4 patients
- Cohort 6; Cohort 7; Cohort 8; Cohort 10: 45mg HB prilocaine following CRM results, 4 patients
- Cohort 9: 40mg HB prilocaine following CRM results, 4 patients
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Statistical analysis (Mean +/- SD) was realized for the total number of patients for each dose proposed by CRM.
Groups:
- Total: Total of all reporting groups
Arm/Group | 35mg HB Prilocaine | 40mg HB Prilocaine | 45mg HB Prilocaine | 50mg HB Prilocaine | Total
Number analyzed (Participants) | 4 | 12 | 20 | 4 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (8.76) | 35.08 (5.11) | 32.85 (4.93) | 29.85 (5.94) | 32.75 (5.69)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4 | 12 | 20 | 4 | 40
  Male | 0 | 0 | 0 | 0 | 0
Length [Mean (Standard Deviation); unit: cm] | 159.5 (4.93) | 164.42 (4.45) | 162.8 (6.26) | 157 (6.16) | 162.38 (5.89)
Weight [Mean (Standard Deviation); unit: kg] | 73 (16.02) | 82.17 (11.93) | 79.78 (11.6) | 84.68 (2.88) | 80.31 (11.62)
Gravity [Mean (Standard Deviation); unit: number of pregnancies] | 3 (1.41) | 2.17 (1.03) | 3.1 (1.98) | 2 (0.96) | 2.70 (1.47)
Parity [Mean (Standard Deviation); unit: number of deliveries] | 1.25 (0.5) | 0.67 (0.49) | 1.3 (1.98) | 0.75 (0.96) | 1.05 (1.47)
Previous Caesarean Section (CS) [Count of Participants; unit: Participants]
  no previous caeserean | 2 | 7 | 10 | 3 | 22
  1 previous caeserean | 2 | 5 | 10 | 1 | 18
Term [Mean (Standard Deviation); unit: weeks] | 38.5 (0.58) | 38.42 (1.08) | 38.40 (0.94) | 38.75 (1.26) | 38.45 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Success of Anesthesia
Description: The nerve blockade will be considered as success when a bilateral T4 level will reach in 15 minutes after intrathecal injection without additional epidural injection needed within 45 minutes peri-operative ; no pain at the skin incision, no pain during 45 minutes after the skin incision
Time Frame: during surgery (average 1 hour)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1; Cohort 6; Cohort 7; Cohort 8; Cohort 10: 45mg
- Cohort 2; Cohort 3; Cohort 9: 40mg
- Cohort 4: 35mg
- Cohort 5: 50mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  Success | 4 | 4 | 4 | 1 | 4 | 4 | 4 | 4 | 3 | 3
  Failure | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1

2. Secondary Outcome: Sensitive Block Duration
Description: Level of Sensory block assessed as loss of sensation to cold, every 2 minutes after spinal anesthesia during 15 minutes, then every 5 minutes until the end of surgery, thereafter, once 30 minutes until total regression of sensory block (T12-S1).
Time Frame: Until complete release of sensory block (T12-S1) (average 4 hours)
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
hours | 2.31 (0.48) | 3.25 (0.50)

3. Secondary Outcome: Sensitive Block at End of Surgery
Description: Level of Sensory block assessed as loss of sensation to cold, every 2 minutes after spinal anesthesia during 15 minutes, then every 5 minutes until the end of surgery, thereafter, once 30 minutes until total regression of sensory block (T12-S1). For this study, dermatome levels are depicted on a scale ranging from 1 to 18. (1 to 12 = T1-T12 thoracic levels; 13 to 17 = L1-L5 lumbar levels; 18 = S1 sacral level)
Time Frame: Until complete release of sensory block (T12-S1) (average 4 hours)
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Median (Standard Deviation); unit: Dermatome level
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Dermatome level | 3.88 (1.59) | 3.00 (0.82)

4. Secondary Outcome: Motor Block Duration
Description: Bromage scale (1 = no motor block; 2 = hip blocked; 3 = hip and knee blocked; and 4 = hip, knee, and ankle blocked) was used to evaluate the motor block every 15 minutes after spinal anaesthesia (T0) and until the end of surgery. Duration was defined from the time of the spinal injection until Bromage scale = 1.
Time Frame: Until complete release of motor block (Bromage scale = 1; average 4 hours)
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
hours | 2.75 (0.45) | 3.50 (0.58)

5. Secondary Outcome: Bromage Motor Block Level at End of Surgery
Description: Bromage scale (1 = no motor block; 2 = hip blocked; 3 = hip and knee blocked; and 4 = hip, knee, and ankle blocked) was used to evaluate the motor block every 15 min after spinal anaesthesia (T0) and until the end of surgery.
Time Frame: Until complete release of motor block (average 4 hours)
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
score on a scale | 3.56 (0.51) | 4.00 (0.00)

6. Secondary Outcome: Newborn Apgar Score
Description: Newborn Apgar score assessed at 1, 5, 10 minutes after baby extraction. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from 0 to 2, then summing up the five values thus obtained. The overall resulting score ranges from 0 to 10 ( 0-3 : severely depressed, 4-6 : Moderately depressed and 7-10 : Excellent condition).
  The five criteria are summarized using words chosen to form an abbreviation (Appearance, Pulse, Grimace, Activity, Respiration).
Time Frame: up to 10 minutes after baby extraction
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
score on a scale
  Apgar at 1 minute | 8.47 (1.84) | 9.00 (0.82)
  Apgar at 5 minutes | 9.63 (0.96) | 9.75 (0.50)
  Apgar at 10 minutes | 9.84 (0.50) | 10 (0)

7. Secondary Outcome: Newborn Methemoglobinemia (MetHb)
Description: Newborn Methemoglobinemia (MetHb) will be assessed at delivery by cordal blood sample, as a routine control, and expressed as a percentage of total hemoglobinemia.
Time Frame: average 1 hour
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Mean (Standard Deviation); unit: percentage of MetHb
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 10 | 1
percentage of MetHb | 1.59 (0.53) | 1.60

8. Secondary Outcome: Number of Participants Needing Vasopressors
Description: Arterial blood pressure will be measured at every 2.5 minute during surgery, then at every 20 minutes in the PACU (Post Anesthesia Care Unit). Vasopressors were given for patients with low blood pressure.
  A low blood pressure is defined as a blood pressure lower than 20% or more than the basal blood pressure (Systolic blood pressure before spinal anesthesia).
Time Frame: during surgery (average 1 hour)
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 15 | 2

9. Secondary Outcome: Number of Participants With Transient Neurologic Symptoms (TNS)
Description: TNS are defined as pain and/or dysesthesia occurred after complete release of sensory block at the gluteal level, at the thighs and at the legs. At Day 0, Day 1, Day 3 and Day 5
Time Frame: up to 5 Days
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Nausea or Vomiting
Description: from 15 minutes after spinal anesthesia and every 4 hours for 24 hours (score 0=no symptoms; 1=symptoms with no treatment necessary; 2=symptoms present and treated)
Time Frame: up to 24 hours after surgery
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 3 | 0

11. Secondary Outcome: Number of Participants With Pruritus
Description: as for outcome 10
Time Frame: Up to 24 hours after surgery
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Urinary Retention
Description: All parturients will be questioned for urinary retention (yes or no)
Time Frame: Up to 24 hours after surgery
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Dizziness
Description: All parturients will be questioned for dizziness (yes or no)
Time Frame: Up to 24 hours after surgery
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 5 | 2

14. Secondary Outcome: Number of Satisfied Participants
Description: Maternal satisfaction (yes or no) will be assessed 1 hour after surgery in the PACU (Post Anesthesia Care Unit)
Time Frame: up to 1 hour after surgery
Population: Secondary outcomes are presented only for doses of 45 and 50mg HB prilocaine, which are the nearest of the final ED95
Measure: Count of Participants; unit: Participants
Arm/Group | 45mg HB Prilocaine | 50mg HB Prilocaine
Number analyzed (Participants) | 19 | 4
Participants | 16 | 4

ADVERSE EVENTS:
Arm/Group | 35mg HB Prilocaine | 40mg HB Prilocaine | 45mg HB Prilocaine | 50mg HB Prilocaine
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/12 | 0/20 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/12 | 0/20 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/12 | 0/20 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes